CLINICAL TRIAL: NCT04173104
Title: Pilot Study of [18F]PARPi PET/MR Imaging in Patients With New and/or Suspected Recurrent Brain Tumors
Brief Title: PET and MRI Imaging of Brain Tumors Using [18F]PARPi
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-311
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor; Brain Cancer
Keywords: Brain cancer; 18FPARPi; PET scan; MRI; Memorial Sloan Kettering Cancer Center; 19-311
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Brain Cancer (Experimental): Participants with new or suspected recurrent brain tumors
  Interventions: Diagnostic Test: PET/MR with [18F]PARPi; Drug: [18F]PARPi

INTERVENTIONS:
Diagnostic Test: PET/MR with [18F]PARPi — One PET/MR study (with up to 3 scan times) with [18F]PARPi
Drug: [18F]PARPi — Injection of <100ug of [18F]PARPi prior to 1 PET/MR

SUMMARY:
This study is to collect data about how 18FPARPi can be used together with PET/positron emission tomography and MRI/magnetic resonance imaging scans to take pictures of brain cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with new or suspected recurrent brain tumors (including suspected recurrent brain tumors showing growth from any preceding scan)
* Age >/= 18 years
* Minimum at least one brain lesion size >/= 1.5cm diameter
* Scheduled to undergo treatment at MSK
* Willingness to sign informed consent
* Able to receive intravenous gadolinium contrast per MSK Department of Radiology guidelines

Exclusion Criteria:

* Any contraindication to 3T MRI (PET/MR scanner is 4.0 Tesla)
* Pregnancy or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-02-05 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
SUVmax measurements | Up to 24 weeks
  [18F]PARPi updtake in lesions will be quantified by standard SUVmax measurements from PET/MR scans

CONTACTS AND LOCATIONS:
Overall Officials: Robert Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org